CLINICAL TRIAL: NCT05120596
Title: An Open-label, Phase I/II Study of T3P-Y058-739, a Genetically-modified Strain of the Bacterium Yersinia Enterocolitica, in Patients With Advanced Solid Tumours
Brief Title: First in Human Study of T3P-Y058-739 (T3P)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: T3 Pharmaceuticals AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T3P1001
Record Dates: First submitted 2021-09-14; First posted 2021-11-15 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced; Solid; Tumor; Cancer; Oncology; Genetically; Bacterium; gene
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: dose-finding, safety, and proof-of-concept study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T3P-Y058-739 Intravenous (IV) (Experimental): Intravenous infusion
  Interventions: Drug: T3P-Y058-739 (IV)
- T3P-Y058-739 Intratumoural (IT) (Experimental): Intratumoural injection
  Interventions: Drug: T3P-Y058-739 (IT)
- T3P-Y058-739 plus pembrolizumab (Experimental): Intravenous infusion
  Interventions: Drug: Pembrolizumab+T3P-Y058-739

INTERVENTIONS:
Drug: Pembrolizumab+T3P-Y058-739 — intravenous infusion or intratumoural injection
  Arms: T3P-Y058-739 plus pembrolizumab
Drug: T3P-Y058-739 (IV) — Intravenous infusion
  Arms: T3P-Y058-739 Intravenous (IV)
Drug: T3P-Y058-739 (IT) — Intratumoral use
  Arms: T3P-Y058-739 Intratumoural (IT)

SUMMARY:
This is a first in human, phase I/II open-label, dose-finding, safety, and proof-of-concept clinical trial of T3P-Y058-739, a genetically-modified, live attenuated strain of the bacterium Yersinia enterocolitica, in patients with advanced solid tumors.

DETAILED DESCRIPTION:
The study, which has a modular design with up to 6 parts, anticipates enrolling approximately 100 participants. Part A will open first. Part B and subsequent parts will open later. The study will evaluate T3P-Y058-739 monotherapy given by intratumoural (IT) injection (Part A) and by intravenous (IV) infusion (Part B). In addition, either IT or IV T3P-Y058-739 (route of administration to be chosen based on emerging data) will be evaluated in combination with pembrolizumab. All patients will receive low doses of desferrioxamine (which provides iron in a form that can be used by the bacteria) to support bacterial survival and growth. All patients will receive antibiotics on completion of therapy to eradicate any residual T3P-Y058-739.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically- or cytologically-proven advanced, unresectable solid tumour for which there is no curative therapy and no alternative therapy is felt to be appropriate.
2. At least one measurable lesion
3. Male or female, 18 years of age or older at the time of signing informed consent.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
5. Estimated life expectancy of ≥12 weeks.
6. Resolution of all acute reversible toxic effects of prior therapy or surgical procedure to baseline or Grade ≤1 (except alopecia).
7. Adequate iron stores without significant iron overload
8. Adequate organ function
9. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF).
10. At least one lesion that is measurable according to iRECIST/RECIST 1.1 and amenable to direct IT injection, i.e., a lesion that is visible, palpable, or detectable by ultrasound, and accessible for direct IT injection (injection via an endoscope is not allowed for Part A at least; ultrasound and/or radiological guidance is allowed).

Exclusion Criteria:

1. Current or prior malignancy that could affect compliance with the protocol or interpretation of results. Patients curatively treated more than 2 years prior to enrolment, and patients with adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ, are generally eligible.
2. Known central nervous system (CNS) metastases.
3. Patients who have previously received an allogeneic bone marrow or stem cell transplant or with congenital or acquired immunodeficiency or receiving immunosuppressive therapy (including any dose of systemic corticosteroids). Patients should have recovered immunologically from any prior immunomodulatory therapies such as CD20-targeted antibodies. Patients receiving inhaled corticosteroids for asthma or chronic obstructive pulmonary disease, and patients on steroid replacement therapy (e.g. due to prior adrenalectomy or hypophysectomy) are eligible at the investigator's discretion. Patients likely to require immunosuppressive treatment with systemic steroids or other agent (e.g., patients with frequent exacerbations of asthma) should not enter the study.
4. Patients with active uncontrolled infection or known to be serologically positive for human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection. Patients with recent major infection (such as pneumonia in the previous 4 weeks) should have recovered to preillness levels with resolution of reversible infection-related symptoms for at least one week prior to starting T3P.
5. Patients with a documented Yersinia infection in the 12 weeks prior to treatment or with detectable Y. enterocolitica in a baseline stool sample (based on routine culture at site).
6. Patients who have recently received antibiotics that could affect the viability of T3P (at least 5 half-lives should have elapsed since the last dose).
7. Patients with known cardiac valvular disease or arterial aneurysms, artificial heart valves and other implanted prostheses (such as joint replacements) that cannot be easily removed or replaced. Patients with central venous access devices are allowed in the study but T3P should be administered by peripheral vein, whenever possible. Patients with a history of bacterial endocarditis, regardless of the organism, are excluded from the study.
8. Patients with a history of clinically significant autoimmune conditions, major cardiac arrhythmia or ischaemia, requiring any form of regular or "as needed" medication to control symptoms, New York Heart Association class II, III or IV cardiac failure or coronary angioplasty in the previous 6 months.
9. Patients who are allergic to chloramphenicol or to all of the following antibiotics: co-trimoxazole, doxycycline, ceftriaxone and cefotaxime.
10. History of hypersensitivity to desferrioxamine
11. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or T3P administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the subject inappropriate for entry into this study. This includes patients on treatment with anticoagulants within 6 months prior to study entry for thromboembolic events.
12. Patients with a bleeding diathesis or receiving therapeutic doses of anticoagulants unless the lesion(s) to be injected are superficial and at low risk of bleeding. Patients receiving lower doses of anticoagulants, aspirin or clopidogrel may be eligible at the investigator's discretion, depending on the site of lesions to be injected and perceived risk of bleeding.
13. Previous severe hypersensitivity reaction to treatment with Check Point Inhibitor (CPI) or other monoclonal antibody.
14. History of severe immune-related adverse effects (irAEs) for greater than 12 weeks. CPI-related AEs (including irAEs) must have resolved back to Grade 0-1 and patients received no corticosteroids for irAEs for at least two weeks prior to first dose of pembrolizumab in the study.
15. History of interstitial lung disease or prior pneumonitis requiring systemic corticosteroid therapy. In case of uncertainty, a high-resolution computed tomography (HRCT) should be performed at baseline.
16. Patients at high risk of bowel perforation, history of acute diverticulitis, intra-abdominal abscess or abdominal carcinomatosis).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-04-26 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Phase 1: To assess the safety and determine the recommended phase II dose (RP2D) when given by IT injection and by IV infusion, as monotherapy and in combination with pembrolizumab. | up to 45 months
  AEs(adverse events), SAEs(serious adverse events) will be graded by the investigator according to National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE Version 5.0).
Phase 2: To assess the safety and preliminary antitumor response T3P when given by IT injection and/or IV infusion, as monotherapy and in combination with pembrolizumab. | up to 45 months
  Response according to immune Response Evaluation Criteria in Solid Tumors (iRECIST) (Seymour et al, 2017).

SECONDARY OUTCOMES:
Assessment of Duration of response (DoR) | up to 45 months
  DoR and PFS according to RECIST 1.1 (Eisenhauer et al, 2009) or modified criteria for selected malignancies, as appropriate(e.g., Verslype et al, 2012 for hepatocellular carcinoma).
Assessment of progression free survival (PFS) | up to 45 months
  PFS according to RECIST 1.1 (Eisenhauer et al, 2009) or modified criteria for selected malignancies, as appropriate(e.g., Verslype et al, 2012 for hepatocellular carcinoma).
To evaluate the distribution of T3P | up to 45 months
  Microbiological culture and/or quantitative polymerase chain reaction (qPCR) of samples of blood, urine, stool and (in patients with tumor's close to or involving the oropharynx) saliva.
To evaluate the clearance of T3P | up to 45 months
  Shedding will also be evaluated in swabs taken from lesions that ulcerate following T3P administration.
To evaluate the shedding of T3P | up to 45 months
  Tumor colonisation will also be evaluated in tumor biopsies (optional).
Assessment of Overall survival (OS) | Maximum 16 months of follow-up
  Overall survival (OS) (maximum 16 months of follow-up).

CONTACTS AND LOCATIONS:
Locations (11):
- Spain (4):
  - Vall d'Hebron Institute of Oncology, Barcelona
  - Institut Catala D'oncologia, L'Hospitalet de Llobregat
  - Hospital Universitario 12 De Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
- Switzerland (3):
  - University Hospital Bern (Inselspital), Bern
  - Centre Hospitalier Universitaire Vaudois Lausanne (CHUV), Lausanne
  - University Hospital of Zürich (Universitätsspital Zürich), Zurich
- United Kingdom (4):
  - Cancer Research UK Clinical trials; Unit Partner in CaCTUS- Cancer clinical trials Unit Scotland; Beatson West of Scotland Cancer Centre, Glasgow
  - Leeds Clinical Research Facility, Leeds
  - Royal Marsden NHS Foundation Trust, London
  - University Hospital Southampton NHS Foundation Trust, Southampton